CLINICAL TRIAL: NCT04291651
Title: Population-Based Analysis of Neoplastic Changes in Cystic Lesions of the Pancreas.
Brief Title: UCSF PANC Cyst Registry
Acronym: UCSF PCR
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 214521
Record Dates: First submitted 2020-02-26; First posted 2020-03-02 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cyst; Pancreatic Neoplasms; Pancreatic Cancer; Pancreatic Diseases; Pancreatic Intraductal Papillary Mucinous Neoplasm; Intraductal Papillary Mucinous Neoplasm; Pancreatic Ductal Adenocarcinoma; Mucinous Cyst
Keywords: Pancreatic Cyst; Pancreatic Cystic Lesion; Pancreatic Cancer; Intraductal Papillary Mucinous Neoplasm; Serous Cystadenoma; Mucinous Cystic Neoplasm; Cancer Epidemiology; Early Detection Research
MeSH Terms: conditions — Pancreatic Cyst; Pancreatic Neoplasms; Pancreatic Diseases; Pancreatic Intraductal Neoplasms; Mucocele; Cystadenoma, Serous | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Patients in this study will have the option of donating blood for biobanking, approximately 10cc of plasma and 10cc of serum. Patients will also have the opportunity to donate a saliva sample at the time of study registration, or at a later date.
  Further, samples that are routinely collected for diagnostic purposes may be collected and banked at the time of their clinically routine procedure. If a patient consents to the use of extra material for research purposes, the biological samples will be banked and the blood, and/or pancreatic juice/cystic fluid, tissues, and saliva will be used for identification and characterization of potential biomarkers from de-identified samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: The registry will be populated with a retrospective cohort of patients previously identified as having pancreatic cysts.
- Prospective: The prospectively enrolled patients in this study are the primary population of interest.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — There are no study-specific interventions, as this is a prospective registry. However, patients will be asked to complete approximately 1-2 hours worth of surveys on things such as demographics, medical and surgical history, and pancreatic cyst-specific questionnaires.
  Groups: Prospective

SUMMARY:
Pancreatic cysts are found incidentally on 15-50% of CT and MRIs for all indications and their prevalence is increasing. Many of these cysts may be precursors to pancreatic cancer, and thus pose a substantial risk, however, the vast majority are benign. Increased detection of pancreatic cysts provides an opportunity to diagnose pancreatic malignancy at an early, curable stage yet also increases the potential to over-treat clinically insignificant lesions. This presents a clinical challenge to prevent unnecessary resection of indolent disease, with associated risks of infections, bleeding, diabetes, and costly disability. Unfortunately, there is little information on the epidemiology and natural history of pancreatic cysts to help guide management.

DETAILED DESCRIPTION:
This study develops a large, prospectively managed, electronic, patient-directed pancreatic cyst registry based at UCSF. The UCSF Pancreatic Cystic Lesions Registry (PANC Cyst) will facilitate work to improve clinical care and understanding of pancreatic cysts by prospective follow-up of patients with cystic lesions, especially the diagnostically challenging small cysts, to identify factors related to cyst formation and progression to malignancy. Longitudinal data capture that includes clinical outcomes will also enable us to more precisely define anatomic, radiographic and biomarker information that can be used to differentiate populations of patients for whom surgery is indicated, surveillance is warranted, or no further evaluation is necessary.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for this study are intentionally broad. Eligible patients for prospective enrollment will include
* Adults ≥ 30 years of age
* Have a radiographic or endoscopic diagnosis of at least one pancreatic cysts regardless of treatment status,
* No history of pancreatic cancer,
* Can speak and read English,
* Have access to a computer or mobile device (~95% of U.S. population); and
* Are able to complete an electronic informed consent.

Exclusion Criteria:

* Patients who don't speak English,
* Don't have access to a computer or mobile device; or
* Patients who have a cancer diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The majority of patients in this study will be over the age of 60 years old, due to the natural age distribution of pancreatic cysts. There will be an approximately even distribution of males and females.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Cancer | 1-10 years
  While not the primary outcome measure, the development of cancer from a pancreatic cyst is a critically important study endpoint, which the investigators do not expect to be frequent occurrence.
Indolency | 1-10 years
  If a patient with a pancreatic cyst experiences no or minimal change in size, and no development of worrisome or high-risk stigmata (Tanaka 2017), this will be considered to be an indolent lesion. Most patients will fall under this category.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly S Kirkwood, MD, Principal Investigator — University of California, San Francisco; Paige M Bracci, PhD, MPH, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No